CLINICAL TRIAL: NCT02285179
Title: Phase I/Prospective Randomized Phase II Trial Of the Safety and Efficacy of Tamoxifen in Combination With GDC-0032 Compared With Tamoxifen alONe.
Brief Title: Clinical Trial to Evaluate the Safety and Effectiveness of GDC-0032 When Given Alongside Tamoxifen
Acronym: Poseidon
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); EurocanPlatform (Unknown); Rather (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M14POS
Record Dates: First submitted 2014-10-21; First posted 2014-11-06 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: GDC-0032; Pi3K inhibitor; tamoxifen; hormone receptor positive; RECIST; pharmacodynamic
MeSH Terms: conditions — Breast Neoplasms | interventions — 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blinded study
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tamoxifen and GDC-0032 (Experimental): 20 mg tamoxifen QD and 4 MG GDC-0032 QOD
  Interventions: Drug: GDC-0032; Drug: Tamoxifen
- tamoxifen and placebo (Placebo Comparator): 20 mg tamoxifen QD and placebo QOD
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: GDC-0032 — Dose of GDC-0032 given orally, once daily (total daily dose) level -1: 2 mg Q.O.D GDC-0032 level 1: (starting) 2 mg QD for 21 days, 7 days off and tamoxifen 20 mg qd level 2: 4 mg QD for 21 days, 7 days off and tamoxifen 20 mg qd
  Arms: tamoxifen and GDC-0032
Drug: Tamoxifen — daily dose of 20 mg

SUMMARY:
This study is designed as a phase 1 dose escalation study followed by a randomised phase II study. The study will be performed in three different centres: Addenbrooke & Cambridge university (Cambridge, UK), Netherlands Cancer Institute Amsterdam), and Vall d'Hebron Hospital (Barcelona, Spain).

Three to six patients will be followed for one completed cycle of therapy (28 days) and subsequent enrolment of new cohorts will be based on the safety assessment in that first cycle and the documentation of dose limiting toxicities. To determine the safety and efficacy of tamoxifen in combination with the isoform selective Pi3K inhibitor GDC-0032 compared with tamoxifen alone.

DETAILED DESCRIPTION:
To determine the recommended phase II dose (RPTD) of GDC-0032 in combination with tamoxifen in hormone receptor positive, HER2 negative metastatic breast cancer patients who have progressed after prior endocrine treatment .Description of toxicity profile, severity and frequency of adverse events (observed with the combination of GDC-0032 and tamoxifen To evaluate the safety and tolerability of GDC-0032 in combination with tamoxifen, recording adverse events using CTCAE v. 4.0 criteria To describe the pharmacokinetics of GDC-0032 in combination with tamoxifen To investigate the possibility of major drug-drug interactions (PK) To obtain proof of target inhibition by selected pharmacodynamic measurements To look for preliminary evidence of anti-tumour activity To assess the status of potential biomarkers for drug response like PIK3CA gene mutations, relevant proteins and phospho-proteins in the PI3K pathway, circulating tumour DNA (ct-DNA) To assess germline DNA sequence for pharmacogenetics studies

ELIGIBILITY:
Inclusion criteria:

Minimum age for inclusion 18 years

* The patient has a WHO performance status ≤ 2
* Premenopausal and postmenopausal female breast cancer patient with histological proven ER and/or PR positive*, HER2 negative breast cancer (based on the most recent assessment of ER and PR status from primary breast cancer or from recurrent or metastatic disease). If a patient is premenopausal by clinical and analytical assessment (defined as having premenopausal follicle stimulating hormone (FSH) and/or plasma estradiol levels), she should also receive a LHRH agonist.
* The patient's breast cancer must be negative for HER2 over-expression by IHC (IHC score ≤1+) or for HER2 gene amplification by FISH or CISH or SISH
* Patients must have either measurable or evaluable disease by RECIST criteria version 1.1.
* The patient has recurrent or metastatic breast cancer that is refractory to an endocrine therapy defined as the occurrence of either of the following while the patient is on endocrine therapy:
* Disease progression of locally advanced or metastatic breast cancer
* Disease recurrence of early stage breast cancer (i.e., recurrence while receiving adjuvant treatment with endocrine therapy)
* Availability of a representative tumour tissue specimen:
* If a patient is currently receiving bisphosphonates, the patient must have received the bisphosphonates for at least 1 month before starting study treatment.
* The patient has adequate organ and marrow function, as defined in protocol.
* The patient has no other diagnosis of malignancy or evidence of other malignancy for 2 years before screening for this study (except non-melanoma skin cancer or in situ carcinoma of the cervix).
* Life expectancy ≥ 12 weeks.
* Fasting glucose ≤ 120 mg/dL (=6.66 mmol/L) and HbA1c ≤ ULN.

exclusion criteria:

* The following restrictions on prior anticancer therapy apply;
* Endocrine therapies or small molecule targeted (non-cytotoxic) inhibitors within 2 weeks or 5 half-lives of the compound or active metabolites, whichever is longer, before the first dose of the study treatment are not allowed

  --No more than 5 prior chemotherapeutic regimens for metastatic breast cancer
* Radiation therapy within 2 weeks before the first dose of study treatment, unless of palliative intent, not compromising bone marrow function
* Cytotoxic chemotherapy within 3 weeks, or nitrosoureas or mitomycin C within 6 weeks before the first dose of the study treatment
* Antibody therapy within 4 weeks before the first dose of the study treatment
* Major surgery or not recovered from major surgery, within 4 weeks before the first dose of study treatment
* Other malignancy with the exclusion of carcinoma in situ.
* The patient has not recovered from toxicity due to prior therapy to grade ≤1 or to pre-therapy baseline. Patients with grade 2 peripheral neuropathy or grade 2 alopecia related to prior therapies are eligible
* The patient has untreated, symptomatic, or progressive brain metastases. -The patient has a history of thrombo-embolic disease or is currently receiving anticoagulation with therapeutic doses of warfarin.
* The patient has prothrombin time/ International Normalized Ratio (PT/ INR) or partial thromboplastin time (PTT) test results at screening that are above 1.3 x the laboratory upper limit of normal.
* Patients with a history of Crohn's disease or ulcerative colitis or other forms of autoimmune colitis
* The patient has uncontrolled significant intercurrent illness
* History of clinically significant cardiac or pulmonary dysfunction-The patient has a type 1 or 2 diabetes requiring daily anti-hyperglycemic medication
* Corticosteroid use equivalent to more than 10mg prednisone daily
* The patient is known to be positive for the human immunodeficiency virus (HIV).
* The patient has a previously identified allergy or hypersensitivity to components of the study treatment formulation(s).
* The patients is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* Pregnant or nursing women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with MTD toxicity | 4 weeks
  MTD toxicity will be assessed in the first 28 days of treatment

SECONDARY OUTCOMES:
Safety Number of patients with adverse events | 2 year
  Number of patients with adverse events
Pharmacokinetics Number of patients with germline DNA sequence | 12 months
  Number of patients with germline DNA sequence
Response Number of patients with a response to protocol treatment | 2 year
  Number of patients with a response to protocol treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sabine C. Linn, prof.dr., Principal Investigator — NKI-AvL; Richard Baird, dr, Study Chair — Cambridge University
Locations (14):
- Gustave Roussy, Paris, France
- Netherlands (6):
  - Antoni van Leeuwenhoek, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Ziekenhuis Groep Twente, Hengelo
  - MUMC, Maastricht
  - Haaglanden Medisch Centrum, The Hague
- Spain (6):
  - Hospital Germans Trias i Pujol, Badalona
  - Vall d'Hebron University Hospital/VHIO, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital ICO-Hospitalet (Bellvitge), Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Universitari Sant Joan de Reus, Tarragona
- University of Cambridge, Cambridge, United Kingdom